CLINICAL TRIAL: NCT03652363
Title: A Placebo-Controlled, Randomised, Double-Blind Trial to Assess the Safety and Efficacy of Intermittent Bilateral Intraputamenal (GDNF) Infusions Administered Via Convection Enhanced Delivery (CED) in Subjects With Parkinson&Apos;s Disease
Brief Title: GDNF in ideopathicParkinsons Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: North Bristol NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2553
Record Dates: First submitted 2018-08-21; First posted 2018-08-29 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Idiopathic Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Glial Cell Line-Derived Neurotrophic Factor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo administered via convection enhanced delivery
  Interventions: Drug: glial cell line-derived neurotrophic factor
- glial derived neurotrophic factor (Experimental): Recombinant-methionyl human glial cell line-derived neurotrophic factor (r-metHuGDNF), administered via convection enhanced delivery
  Interventions: Drug: glial cell line-derived neurotrophic factor

INTERVENTIONS:
Drug: glial cell line-derived neurotrophic factor — Intermittent Bilateral Intraputamenal Glial Cell Line-Derived Neurotrophic Factor (GDNF) Infusions Administered via Convection Enhanced Delivery
  Other Names: GDNF

SUMMARY:
A Placebo Controlled Randomised Trial of GDNF vs placebo

The study will require patients to undergo surgery to implant microcatheters precisely into the brain. Patients will then attend clinic on a 2 weekly basis for infusions of a nerve growth factor called GDNF or placebo. Specific tests will also be carried out at regular intervals to assess your symptoms. All participants will undergo radio-isotope brain imaging at the beginning and end of the study. Periodically patients will also be required to undergo an MRI scan to assess the delivery of the study drug or placebo.

DETAILED DESCRIPTION:
Patients who are considered likely to meet certain suitability criteria for this trial and who provide fully informed consent to participate will have screening blood tests and clinical assessments. As part of these assessments patients will be asked to stop their PD medication overnight to allow us to assess the severity of their PD symptoms without the benefit of medication on board. These assessments will answer if patients are eligible to enter the trial. Some patients will not continue on with the trial following these assessments. However, we will discuss with those patients alternative clinical care / research options.

Patients that are felt to be eligible for the trial following these assessments will undergo brain surgery performed under general anaesthetic. During the surgery 4 tiny plastic infusion tubes will be inserted into the putamen area of the brain, 2 on either side of the brain (two in each putamen). These tubes connect to a single metal port that will come out (exit) from under the skin behind the ear. This port can be accessed as needed from the outside and will allow GDNF or placebo infusions to be given every 4 weeks directly into the putamen part of the brain without requiring additional surgery or piercing of the skin (see Figure 1).

Approximately 4 weeks after surgery patients will have an infusion of placebo / dummy drug and an MRI to check the tubes and port system are working well enough to allow infusions of either GDNF or placebo (further details below).

Patients will be required to attend NBT in order to have either GDNF or placebo infusions given through the port and down the tiny plastic tubes into the putamen every 4 weeks for a total of 9 months (10

infusions in total). Neither the patient nor the research team will know whether patients are receiving GDNF or placebo / dummy infusions.

For some of these visits, patients will again be asked to stop their PD medication the night before. By doing this, it will be possible to assess potential reversal of symptoms compared with before the start of brain infusion treatments.During the course of this trial patients will undergo positron emission tomography (PET) brain scans at another hospital on two or three occasions to look for evidence of damaged brain cell recovery. This trial is therefore time-consuming and this will be made clear to you before seeking your consent to participate.

We hope that this trial will help clarify whether GDNF does indeed have the potential to reverse Parkinson's disease and restore parts of the brain. It must be understood, however, that even if the trial yields positive results, further testing will be required in a larger number of patients to meet the requirements of the health authorities prior to GDNF being available over the long term or routinely.

Participation in this trial will involve some risks to patients. These risks are described in detail later in this document and will be discussed with you before you give informed consent. When the trial ends the information collected from participants will be used to produce reports for scientific journals, and will be presented at scientific meetings so that doctors and scientists around the world will better understand the potential brain restoring and disease reversing effects of GDNF in PD.

ELIGIBILITY:
Inclusion Criteria:

In order to qualify for entry into the presurgery and surgery and healing periods of the study, subjects MUST meet all of the following criteria:

1. Subjects diagnosed with idiopathic PD according to the United Kingdom (UK) Brain Bank Criteria. Bilateral findings must be present at study entry.
2. Duration of PD ≥ 5 years.
3. Age 35-75 years.
4. Presence of motor fluctuations. Subjects must have an average of at least 2.5 hours of OFF-time per day on 3-day fluctuation diaries completed during screening.
5. Ability to reliably distinguish motor states (ON without dyskinesias, ON with non-troublesome dyskinesias, ON with troublesome dyskinesias and OFF) and accurately complete fluctuation diaries.
6. UPDRS motor score (part III) in a practically defined OFF-state between 25-45.
7. Hoehn and Yahr ≤ stage III in the OFF-state.
8. Responsiveness to levodopa (> 40% improvement in motor UPDRS [part III] following a levodopa challenge).
9. No change in anti-parkinsonian medication for 6 weeks before screening.
10. Females of childbearing potential must have a negative pregnancy test at study entry and be willing to use an approved (by the PI or designee) form of contraception until the end of the study.
11. Provision of informed consent. -

Exclusion Criteria:

Subjects who meet any of the following criteria will NOT be eligible for entry into presurgery and surgery and healing periods of the study:

1. Diagnosed with atypical parkinsonism or any known secondary parkinsonian syndrome including but not limited to medication induced, toxic, vascular, post-traumatic or post-infectious parkinsonism, progressive supranuclear palsy, multiple systems atrophy, or other neurodegenerative disorder associated with parkinsonism.
2. Signs or symptoms suggestive of atypical parkinsonian syndrome including supranuclear gaze palsy, early postural instability and falls (within 3 years of disease onset), cerebellar signs, myoclonus, disproportionate antecollis, extensor plantar responses, cortical sensory loss, emotional incontinence (pseudobulbar affect), severe bulbar dysfunction (dysarthria, dysphonia or dysphagia) or respiratory symptoms such as stridor or inspiratory sighs.
3. Family history of more than 1 first-degree relative with PD.
4. Severe dyskinesias or severe tremor which could interfere with GDNF infusion.
5. Prior neurosurgical treatment for PD, including previous treatment with GDNF or deep brain stimulation.
6. Significant neurological disorder other than PD including clinically significant head trauma, cerebrovascular disease, CSF shunt or other implanted CNS device.
7. Presence of significant depression as defined as a Beck Depression Inventory (BDI) score ≥ 14.
8. Current or past history of psychosis requiring therapy. The presence of benign hallucinosis is not exclusionary.
9. Presence or history of clinically significant impulse control disorder or presence or history of dopamine dysregulation syndrome.
10. MoCA score < 24.
11. Use within 3 months of planned catheter insertion of concomitant medications known to affect PD symptoms other than prescribed PD therapy including but not limited to neuroleptics or other central dopamine receptor blockers.
12. Any medical condition which might impair outcome measure assessments or safety measures including ability to undergo MRI scanning.
13. Screening MRI demonstrating any abnormality which would suggest an alternative cause for subject's parkinsonism.
14. Any medical condition that would put the subject at undue risk from surgical treatment or chronic implants including but not limited to bleeding disorders, chronic infections, or immunosuppressive illness.
15. History within the last 5 years of cancer with the exception of basal cell carcinoma of the skin.
16. History of drug or alcohol abuse within 2 years of planned catheter insertion.
17. Use of any investigational drug or device within 90 days of planned catheter insertion.
18. Active breastfeeding. 5.3.4 Post-Surgery Randomisation Criteria

In order to be eligible for entry into the double-blind period of the study, subjects must meet the following criteria after undergoing surgery:

1. No relevant sequelae from catheter implantation such as clinically significant intracerebral trauma, haemorrhage, or infection.
2. Total distribution volume providing at least 50% volume coverage of a predefined volume of interest in each putamen (approximately 25% volume coverage of total putamen), as assessed by an independent review of an MRI scan taken within 2 hours post-infusion of diluent at the end of the healing period.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2012-10-25 (Actual); Primary Completion 2015-03-13 (Actual); Study Completion 2016-04-01 (Actual)

PRIMARY OUTCOMES:
UPDRS in the off state | 40 weeks
  The primary outcome for this study will be the percentage change in motor UPDRS in the practically defined OFF state between baseline and Week 40.